CLINICAL TRIAL: NCT04168346
Title: Preoperative Intravenous Iron Therapy in Patients With Gastric Cancer
Acronym: IRONSTOMACH
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Ville Sallinen, MD, Phd, Adj. Professor, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HUS/333/2019
Record Dates: First submitted 2019-11-12; First posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Gastric Cancer; Anemia; Surgery; Iron Deficiency Anemia; Surgery--Complications
MeSH Terms: conditions — Stomach Neoplasms; Anemia; Anemia, Iron-Deficiency | interventions — ferric carboxymaltose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): IV-iron substitution: The intravenous iron formulation used in the study is ferric carboxymaltose and it will be administered two to four weeks before the surgery, aiming at four weeks. The dose of intravenous iron will be calculated according to the weight and haemoglobin level of the patients, however so that all the patients receive minimum 1000mg iv iron and the maximum dose is 20 mg/kg per day.
  Interventions: Drug: Ferric carboxymaltose
- Placebo (Placebo Comparator): Placebo is NaCl 0.9% solution, which is administrated in the same way as the study drug
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Ferric carboxymaltose — Ferric carboxymaltose iv infusion
  Arms: Intervention
Drug: Placebos — NaCl 0.9% infusion
  Arms: Placebo

SUMMARY:
The main objective of this investigator initiated study is to study if preoperative intravenous iron is effective in reducing need for allogenic blood transfusion in patients with gastric cancer who will undergo a standardized gastrectomy including both total and subtotal gastrectomies. The hypothesis is that intravenous iron reduces the need for perioperative blood transfusions.

ELIGIBILITY:
Inclusion Criteria:

- Patients with gastric cancer who will undergo a gastrectomy

Exclusion Criteria:

* Patients under 18 years old
* Patients not in full understanding
* Hemoglobin levels > 155 g/l for women and >167 g/l for men (upper reference limits for the laboratory of Helsinki University Hospital district) preoperatively.
* Transferrin saturation level >50%
* Emergency gastrectomy
* Palliative gastrectomy
* Acute bacterial infection
* Known hypersensitivity to the active substance, to ferric carboxymaltose or any of its excipients, or to other parental iron products
* Clinical evidence of iron overload or disturbances in the utilisation of iron
* Patients <35 kg
* Dialysis therapy for chronic renal failure
* Hemochromatosis
* Polycythemia vera
* Pregnancy
* Patients in need of direct blood transfusion ( Criteria for this are hemoglobin < 80 g/l or < 90 g/l if the patient is symptomatic or has a history of heart disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
The need for blood transfusion | Within 30 days from the day of the operation
  Number of patients needing transfusions

SECONDARY OUTCOMES:
Postoperative complications | Within 30 days from operation
  Postoperative complications measured using Comprehensive complication index
Patients' quality of life (RAND) | One and six months after the surgery
  RAND questionnaires
Patients' quality of life (15D) | One and six months after the surgery
  15D questionnaires
Patients' quality of life (EQ-5D) | One and six months after the surgery
  EQ-5D questionnaires
Patients' quality of life (FRAIL) | One and six months after the surgery
  FRAIL questionnaires
Patients' quality of life (PRISMA-7) | One and six months after the surgery
  PRISMA-7 questionnaires
Patients' quality of life (GSRS) | One and six months after the surgery
  GSRS questionnaires
Patients' quality of life (IDQ) | One and six months after the surgery
  IDQ questionnaires
Patients' haemoglobin and iron parameter levels | At the time of hospital discharge (estimated on average 10 days after surgery)
  Patients' haemoglobin and iron parameter levels
Patients' haemoglobin and iron parameter levels | One month after the surgery
  Patients' haemoglobin and iron parameter levels
Patients' haemoglobin and iron parameter levels | Three months after the surgery
  Patients' haemoglobin and iron parameter levels
Re-admission | 30 days after discharge from hospital
  Patient re-admission rates
90-day mortality | Within 90 days from operation
  90-day mortality
Overall survival | 1, 3 and 5 years from operation
  Overall survival
Length of hospital stay | Within hospital stay, on average 7 - 14 days
  Length of hospital stay
Use of IV iron after operation | Within 3 months from operation
  Number of doses and median dose of IV iron

CONTACTS AND LOCATIONS:
Overall Officials: Arto Kokkola, MD, Study Director — Helsinki University Central Hospital

IPD SHARING:
Plan to Share IPD: No